CLINICAL TRIAL: NCT03353766
Title: The Effect of Timing on Lateral Crossbite Correction - a Randomized Study
Brief Title: Early Crossbite Correction - a Randomized Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oulu (Other)
Collaborators: Oulu University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EETTMK:124/2008
Record Dates: First submitted 2016-08-08; First posted 2017-11-27 (Actual); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Malocclusion; Crossbite
Keywords: Early Orthodontic treatment; Orthodontic treatment outcome; Crossbite treatment
MeSH Terms: conditions — Malocclusion | interventions — Palatal Expansion Technique

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early crossbite correction (Experimental): Early crossbite correction with Q-H Device
  Interventions: Device: Early crossbite correction with Q-H Device
- Crossbite correction in mixed dentition (No Intervention): Later crossbite correction, during mixed dentition

INTERVENTIONS:
Device: Early crossbite correction with Q-H Device — Crossbite treatment in deciduous dentition with Quad-Helix appliance
  Other Names: Expanding device, Maxillary expansion
  Arms: Early crossbite correction

SUMMARY:
The aim of this longitudinal randomized investigation is to determine the long-term effects of early lateral crossbite correction with Quad-Helix appliance, during the deciduous dentition, on craniofacial structures and dental arches, compared to treatment started later, after the first permanent molars have erupted.

The hypothesis is that the timing of treatment has significant effects on orthodontic treatment total time, the general outcome of the treatment, and the compliance of the patient.

The Age cohort of five-year-old of children living in the community areas of Oulunsalo are screened at the age of 5 years for malocclusions. Of these children 80 children who meet the criteria are chosen for the study after the written consent.

The children are randomized into two groups. In the first group the treatment with Quad-Helix appliance is started at the age of 5 to 6 years, before the eruption of the permanent molars. The device is cemented to the second deciduous molars. The treatment is continued and continued until normal lateral occlusion is achieved and the device is kept stable for one year after this.

In the second group headgear treatment is started after the first permanent maxillary molars have erupted. The device is cemented to the first permanent molars. The treatment is continued until normal lateral occlusion is achieved and the device is kept stable for one year after this.

In both groups dental casts, cephalograms, and standardized 3D facial photographs are taken before treatment (T0), after the first treatment phase (T1), after the second treatment phase (T2) and after the growth (T3).

Facial 3D scanning is performed for all the subjects after the treatment to find out the effect of different treatment methods on facial characteristics. The dental casts are scanned to make 3D models of the cast to be used in detailed analysis.

A wide multi-level questionnaire is performed before, during and after the study to the parents and the children to find out the comprehensive effects of orthodontic treatment on the well-being of the child. The questionnaire includes the Rutter's child behavioural pattern (Rutter et al., 2001).

In both studies, all the guidelines of RCT are applied. Blinding of the clinicians is gained, as the orthodontists or dentists treating the children are not aware of the rationale of the study. Blinding is applied on all measurement of the documents.

DETAILED DESCRIPTION:
1. The aim of this longitudinal randomized investigation is to determine the long-term effects of early lateral crossbite correction with Quad-Helix appliance, during the deciduous dentition, on craniofacial structures and dental arches, compared to treatment started later, after the first permanent molars have erupted.
2. The aim was further to find out the possible benefits and the burden of early treatment to the patients and parents of these common malocclusions, when compared to groups treated later, but with the same methods as much as possible.
3. The hypothesis is that the timing of treatment has significant effects on orthodontic treatment total time, the general outcome of the treatment, and the compliance of the patient.
4. Background. In spite of the fact that about 30 to 50% of the children in Europe undergo orthodontic treatment during growth, negligible amount of RCT based data is available concerning these treatments.
5. The most used treatment method in Finland, and one of the most popular in the world, is to treat lateral malocclusion with the maxillary dental arch expanding Quad-Helix appliance (Bodoy et al., 2011; Petren et al., 2011; Lippold et al., 2013).

   The goal of the expansion treatment is typically described as to expand maxillary dental arch, expand the maxilla and correct the possible functional shift in the occlusion.

   The views of the effects of the expanding devices during early childhood are to some extent inconclusive, at least when the long-term effects are concerned. Most reports that are based on a short-term follow-up, describing maxillary arch expansion and the correction of the crossbite. When the Quad-Helix appliance is compared to the removable appliance, the Q-H is found to be more effective (Petren et al., 2011). When it comes to the elimination of the functional lateral shift after the crossbite treatment, the research data is weak and not sufficient (Tsanidis et al., 2016). Valid evidence based data is rare and the thus exact conclusions are very difficult to be set.
6. Preliminary Studies. The investigators conducted a randomized clinical study with an expanding Headgear device, where the control group was treated with a camouflage treatment, without expansion in the adolescence. The main difference between the groups was broader dental arch with less extractions in the headgear group, the differences between the groups being relatively small, except the broader dental arch in the Headgear group. (Mäntysaari et al.,2004; Pirttiniemi et al.,2005; Krusinskiene et al., 2008). However, canine eruption pattern was found to be more favorable in the early headgear group (Silvola et al., 2008).
7. Experimental Design and Methods

   * The Age cohort of five-year-old of children living in the community areas of Oulunsalo are screened at the age of 5 years for malocclusions. Of these children 80 children who meet the criteria are chosen for the study after the written consent. The inclusion criteria are crossbite of at least two deciduous lateral teeth.
   * Exclusion criteria are anterior crossbite, missing permanent teeth, or craniofacial anomaly.
   * The subjects are randomized into two groups. In the first group the treatment with Quad-Helix appliance is started at the age of 5 to 6 years, before the eruption of the permanent molars. The device is cemented to the second deciduous molars. The treatment is continued and continued until normal lateral occlusion is achieved and the device is kept stable for one year after this.
   * In the second group headgear treatment is started after the first permanent maxillary molars have erupted. The device is cemented to the first permanent molars. The treatment is continued until normal lateral occlusion is achieved and the device is kept stable for one year after this In both groups dental casts, cephalograms, and standardized 3D facial photographs are taken before treatment (T0), after the first treatment phase (T1), after the second treatment phase (T2) and after the growth (T3).

   Facial 3D scanning is performed for all the subjects after the treatment to find out the effect of different treatment methods on facial characteristics. The dental casts are scanned to make 3D models of the cast to be used in detailed analysis.
   * A wide multi-level questionnaire is performed before, during and after the study to the parents and the children to find out the comprehensive effects of orthodontic treatment on the well-being of the child. The questionnaire includes the Rutter's child behavioral pattern (Rutter et al., 2001).
   * In both studies, all the guidelines of RCT are applied (Moher and Schulz, 2005). Blinding of the clinicians is gained, as the orthodontists or dentists treating the children are not aware of the rationale of the study. Blinding is applied on all measurement of the documents.
8. Quality assurance plan. Quality of the data collected is secured by preliminary training that has been done concerning the input data and the registration processes. The collected data is monitored on regular basis, on clinical records this is done by three months intervals. The quality assurance of the clinical data is done by the same person who has trained the dental personnel by on-site monitoring and auditing. Immediate feed-back is given to the registering personnel concerning the quality of the records.

   The input data is monitored by testing the normality of the data during the input process. Immediate feed-back is given to the personnel doing the registration process in the cases of deviation is found in the range of normality or consistence of the data. Basic assumption is that the input data is supposed to be normally distributed with this type of patient material.

   Intra- and Inter-examiner error is tested during the measuring process to test the accuracy of the measurements. The level of error is compared to the level of level reached in corresponding studies.
9. Sample size assessment Power and sample size calculation has been made using the data derived from the preliminary studies (Mäntysaari et al., 2004), and the applied sample size was gained using the formula for the purpose:(http://stat.ubc.ca/~rollin/stats/ssize/n2.html).

   The used estimates for means and deviations were gained from the analogous preliminary study. The test power used in the power analysis was 0.80 with the level of significance p=0.05. The used value give the sample size 49, and thus the used sample is very sufficient.
10. Plan for missing data. It is known from earlier longitudinal orthodontic studies that the drop-out rate is about 20% when reaching the end point of the study. This has been taken into account in the original sample size. As randomization is applied, it is likely that the missing subjects will occur approximately at the same rate in both study groups and by choosing appropriate statistical methods, the data can be handled.
11. Statistical analysis plan. The study hypothesis is tested by using statistical methods. When the differences between the two groups are tested, a test for two independent samples is utilized. When the values of the children are compared at different time points, a test of related samples is used. If the sample data is not normally distributed, a non-parametric test is applied ( e.g. Mann-Whitney-test or Wilcoxon-test). When the behavioral items are tested, the applied tests are on ordinary level or nominal level (e.g. Cross-tabulation tests).

    To estimate the Intra-examiner and Inter-examiner error, double measurements are performed. The statistical testing of the error is done using Intra class correlation (ICC).

    The Intention to treat principle is applied in the study. The results will be shown both in graphical and table format to clearly show group and individual variation. The statistical testing is done by using the latest version of SPSS program.
12. Timing and Importance of the studies The first part of the study will be initiated in 2016. The study will continue actively during the years 2016-2019.

The treatments and the follow-up continues until the growth is over, until about year 2028, and further until the adulthood. Most of the data, however, is available to be analyzed already earlier in 2018-2020.

The results of these studies are clinically very important and therefore they will be published in the most respected international orthodontic journals. As the results are of the highest clinical relevance with a sound evidence, they can easily be applied directly to clinical practices.

University of Oulu will give all the facilities needed for the research, including rooms. The clinical examinations are performed in the health centers as a part of normal treatment costs, when normal documentation is concerned.

ELIGIBILITY:
Inclusion Criteria:

* Crossbite of at least two deciduous lateral teeth
* Full deciduous dentition
* Age 5 to 6 years

Exclusion Criteria:

* Anterior crossbite
* Missing permanent teeth,
* Craniofacial syndrome, Cleft lip/palate

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-04; Primary Completion 2021-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Normal occlusion, no lateral crossbite, normal measured Overjet and Overbite | 13 years
  Normal occlusion is measured as:
  * harmonous occlusal contacts, no lateral crossbite
  * Overbite 1 mm to 4 mm
  * Overjet 1mm to 4 mm

SECONDARY OUTCOMES:
Patient compliance, questionnaire | 6 years
  Eariler tested questionnaire is used to compare compliance a different treatment ages
Stability of occlusion in long-term follow-ups. | 13 years
  Normal occlusion, no lateral crossbite, Normal measured Overbite and Overjet in mm
  * Overbite 1 mm to 4 mm
  * Overjet 1mm to 4 mm

OTHER OUTCOMES:
Measured degree of facial asymmetries | 13 years
  * Facial asymmetry measured on 3D photographs in lower facial area in%
  * Facial asymmetry measured on 3D phptpgraphs in middle facial area in%

CONTACTS AND LOCATIONS:
Overall Officials: Anna-Sofia Silvola, Dr., Principal Investigator — University of Oulu
Locations (1):
- University of Oulu, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No
At the moment there is no such plan

REFERENCES:
- [Background] Krusinskiene V, Kiuttu P, Julku J, Silvola AS, Kantomaa T, Pirttiniemi P. A randomized controlled study of early headgear treatment on occlusal stability--a 13 year follow-up. Eur J Orthod. 2008 Aug;30(4):418-24. doi: 10.1093/ejo/cjn021. Epub 2008 Jul 16. PMID 18632838
- [Background] Lippold C, Stamm T, Meyer U, Vegh A, Moiseenko T, Danesh G. Early treatment of posterior crossbite--a randomised clinical trial. Trials. 2013 Jan 22;14:20. doi: 10.1186/1745-6215-14-20. PMID 23339736
- [Background] Mantysaari R, Kantomaa T, Pirttiniemi P, Pykalainen A. The effects of early headgear treatment on dental arches and craniofacial morphology: a report of a 2 year randomized study. Eur J Orthod. 2004 Feb;26(1):59-64. doi: 10.1093/ejo/26.1.59. PMID 14994883
- [Background] Petren S, Bjerklin K, Bondemark L. Stability of unilateral posterior crossbite correction in the mixed dentition: a randomized clinical trial with a 3-year follow-up. Am J Orthod Dentofacial Orthop. 2011 Jan;139(1):e73-81. doi: 10.1016/j.ajodo.2010.06.018. PMID 21195260
- [Background] Pirttiniemi P, Kantomaa T, Mantysaari R, Pykalainen A, Krusinskiene V, Laitala T, Karikko J. The effects of early headgear treatment on dental arches and craniofacial morphology: an 8 year report of a randomized study. Eur J Orthod. 2005 Oct;27(5):429-36. doi: 10.1093/ejo/cji025. Epub 2005 Jun 16. PMID 15961567
- [Background] Silvola AS, Arvonen P, Julku J, Lahdesmaki R, Kantomaa T, Pirttiniemi P. Early headgear effects on the eruption pattern of the maxillary canines. Angle Orthod. 2009 May;79(3):540-5. doi: 10.2319/021108-83.1. PMID 19413375
- [Background] Tsanidis N, Antonarakis GS, Kiliaridis S. Functional changes after early treatment of unilateral posterior cross-bite associated with mandibular shift: a systematic review. J Oral Rehabil. 2016 Jan;43(1):59-68. doi: 10.1111/joor.12335. Epub 2015 Aug 8. PMID 26257271
- [Result] Godoy F, Godoy-Bezerra J, Rosenblatt A. Treatment of posterior crossbite comparing 2 appliances: a community-based trial. Am J Orthod Dentofacial Orthop. 2011 Jan;139(1):e45-52. doi: 10.1016/j.ajodo.2010.06.017. PMID 21195256